CLINICAL TRIAL: NCT01881074
Title: The Influence of Periodontal Treatment on Gingival Inflammatory Response of the Type II Diabetic Patient
Brief Title: Periodontal Treatment Response in Type II Diabetic Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Other Study IDs: 287-2011; CRO-2011-PERIO-01-FP (Other: Colgate-Palmolive)
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Type II Diabetes; Periodontal Disease
Keywords: Type II Diabetes; Periodontal Disease; Periodontitis; Gum Disease; Gingivitis; Triclosan; Inflammatory Markers; Immune Response
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases; Periodontitis; Gingival Diseases; Gingivitis | interventions — hydrated silica gel-based toothpaste; Sodium Fluoride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, gingival crevicular fluid, and saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Triclosan containing toothpaste: Patients with type II diabetes will receive triclosan containing toothpaste and will be asked to brush their teeth using only this toothpaste for the duration of the study (12 months). Patients will be asked to return for an oral exam, dental cleaning and sample collection for up to 12 months following their baseline appointment.
  Interventions: Drug: Triclosan containing toothpaste
- Non-triclosan containing toothpaste: Patients with type II diabetes will receive non-triclosan containing toothpaste and will be asked to brush their teeth using only this toothpaste for the duration of the study (12 months). Patients will be asked to return for an oral exam, dental cleaning and sample collection for up to 12 months following their baseline appointment.
  Interventions: Drug: Non-triclosan containing toothpaste

INTERVENTIONS:
Drug: Triclosan containing toothpaste — Type II diabetic patients will be instructed to brush their teeth at the same time day and with the same frequency as usual for them using only the triclosan containing toothpaste provided to them. Additional tubes of triclosan containing toothpaste will be provided to the participants for the duration of the study as needed. Following their baseline appointment, patients will be asked to return at 6 weeks, 3, 6, 9 and 12 months for an oral exam and dental cleaning. Samples will be collected at baseline, 3, 6 and 12 months. Samples collected may include venous blood, gingival crevicular fluid, plaque and saliva. Female study participants may be asked to perform a pregnancy test.
  Other Names: Colgate Total
  Groups: Triclosan containing toothpaste
Drug: Non-triclosan containing toothpaste — Type II diabetic patients will be instructed to brush their teeth at the same time day and with the same frequency as usual for them using only the non-triclosan containing toothpaste (i.e. placebo) provided to them. Additional tubes of non-triclosan containing toothpaste will be provided to the participants for the duration of the study as needed. Following their baseline appointment, patients will be asked to return at 6 weeks, 3, 6, 9 and 12 months for an oral exam and dental cleaning. Samples will be collected at baseline, 3, 6 and 12 months. Samples collected may include venous blood, gingival crevicular fluid, plaque and saliva. Female study participants may be asked to perform a pregnancy test.
  Other Names: Colgate
  Groups: Non-triclosan containing toothpaste

SUMMARY:
Diabetes mellitus affects > 171 million people worldwide, with type II diabetes being the most prevalent, affecting 85-95% of the diabetic population. Unfortunately, despite conventional medical treatment, some diabetic patients do not seem to be able to reach desirable metabolic control. This is a double-blinded, randomized study investigating the effects of triclosan containing toothpaste (commercial name: Colgate Total) on the response to periodontal treatment in type II diabetic patients with periodontal disease. The investigators believe that using triclosan containing toothpaste during periodontal treatment will decrease the local inflammatory response and that this reduction will improve periodontal status and metabolic control.

DETAILED DESCRIPTION:
Many studies have shown a relationship between chronic inflammatory periodontal diseases and diabetes, in which both diseases influence the other. Research studies have shown that controlling inflammation of the gums can improve the level of metabolic control (i.e. blood glucose levels) in patients with diabetes. However, it is still not clear which periodontal treatment approach would best maintain the control of inflammation of diabetic patients. Triclosan has anti-plaque and anti-inflammatory properties and decreases gum inflammation. The purpose of this study is to 1) determine the effects of triclosan containing toothpaste on gum inflammation in type II diabetic patients with periodontal disease, and 2) to evaluate whether type II diabetic patients will show improvement in periodontal status and blood glucose following periodontal treatment with and without the use of a triclosan containing toothpaste.

Patients with type II diabetes that meet the study criteria will be randomly assigned either triclosan containing toothpaste or placebo toothpaste. Dental cleanings and oral exams will be performed at baseline, 6 weeks, 3, 6, 9 and 12 months, and samples will be collected at baseline, 3, 6 and 12 months. Samples that may be collected include blood, plaque, gingival crevicular fluid, saliva and plaque. Women may also be asked to complete a pregnancy test. Photographs and x-rays of the patients mouth/teeth may be taken, but is not a requirement.

The samples collected will be used to assess the effect of triclosan containing toothpaste on glycemic control and local and systemic inflammatory mediators during the course of periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject males or females 18 to 70 years old
* Subject able and willing to follow study procedures and instructions
* Subject read, understood and signed an informed consent form
* Subject diagnosed with type II diabetes
* Currently under standard treatment and physicians care for diabetes control
* Standard diabetes medication has not changed in the last 3 months
* HbA1c levels of ≥ 6.5% determined upon medical record review within the last 6 months (if HbA1c value not available in medical record or if patient is new, the first study visit value will determine if patient may continue in the study)

Exclusion Criteria:

* Subject with concomitant periodontal therapy 6 months prior to enrollment
* Subject with orthodontic appliances
* Subject chronically treated (i.e., two weeks or more) with any medication known to affect inflammation or periodontal status or (e.g.phenytoin, cyclosporine, Coumadin or steroids) within one month of the first examination*
* Subject currently smoke or who report smoking within one year of first examination ≥ 10 cigarettes/day
* Subject treated with antibiotics within 3 months prior to enrollment
* Subject necessitating antibiotic prophylaxis
* Female subject who report being pregnant or lactating at first appointment
* Subject uses hormonal contraceptives but started method less than 30 days prior to the first examination
* Subject with active infectious diseases (hepatitis, human immunodeficiency virus or Tuberculosis) or subject is immunocompromised as determined by the Investigator
* Subjects has a medical condition which precludes not eating/drinking for approximately 8 hours
* Subject has serious diabetic complications such as macrovascular diseases or kidney or liver failure
* Subjects who have a known allergy to oral care products or ingredients in oral care products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type II diabetic patients with periodontal disease requiring periodontal treatment.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Periodontal Parameters | Baseline, 3, 6 and 12 months
  The changes in clinical parameters(i.e. pocket depth, plaque, clinical attachment loss) during periodontal treatment from baseline to 3 months, 6 months and 12 months. Clinical parameters will be assessed using a conventional periodontal probe and recorded in supporting software (Florida Probe).
Local Inflammatory Markers | Baseline, 3, 6 and 12 months
  The changes in local inflammatory markers (i.e. cytokines, chemokines, metalloproteinases) during periodontal treatment from baseline to 3 months, 6 months and 12 months. Local inflammatory markers in gingival crevicular fluid will be assayed in the laboratory.

SECONDARY OUTCOMES:
Glycemic Control | Baseline, 3, 6 and 12 months
  The changes in glycemic control (i.e. HbA1C levels) during periodontal treatment from baseline to 3 months, 6 months and 12 months. Blood will be analyzed by the core lab facility at the University of Florida and Shands hospital and in the clinic/laboratory using a commercially available finger prick device and testing strips.
Systemic Inflammatory Markers | Baseline, 3, 6 and 12 months
  The changes in systemic inflammatory markers (i.e. cytokines, chemokines, metalloproteinases) during periodontal treatment from baseline to 3 months, 6 months and 12 months of periodontal treatment. Inflammatory markers in venous blood will be assayed in the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana M Shaddox, DDS, MS, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Tokatlian J, Al-Sabbagh M, Dawson DR, Pearce KA, Andriankaja MO, Adatorwovor R, Miguel MMV, Shaddox LM. The impact of periodontal therapy on clinical and inflammatory parameters in type II diabetics. J Periodontol. 2026 Jan 19. doi: 10.1002/jper.70035. Online ahead of print. PMID 41553854